CLINICAL TRIAL: NCT02808897
Title: Active Clearance of Chest Tubes After Cardiac Surgery: A Prospective Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: ClearFlow, Inc. (Industry); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MP-33-2015-1901
Record Dates: First submitted 2016-06-14; First posted 2016-06-22 (Estimated); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation; Pericardial Effusion; Pleural Effusion; Hemothorax; Cardiac Tamponade
Keywords: Chest tubes; Atrial fibrillation; Thoracic surgery; Critical care
MeSH Terms: conditions — Atrial Fibrillation; Pericardial Effusion; Pleural Effusion; Hemothorax; Cardiac Tamponade

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard drainage (Active Comparator): The control arm consist of consecutively enrolled cardiac surgery patients receiving one standard chest tube in the mediastinum and at most three (3) commercially available standard or silastic chest tubes in the mediastinal, right or left pleural space.
  Interventions: Device: Standard drainage
- Active Tube Clearance drainage (Experimental): The test arm consists of consecutively enrolled cardiac surgery patients receiving one (1) chest tube using active tube clearance (PleuraFlow®) in the mediastinum and at most three (3) other commercially available standard or silastic chest tubes in the mediastinal, right or left pleural space.
  Interventions: Device: Active Tube Clearance drainage

INTERVENTIONS:
Device: Standard drainage — One (1) chest tube must be placed in the anterior mediastinum. The other chest tube(s) may be placed at the discretion of the operator. Chest tubes with internal diameter 28 French (Fr) shall be used. Use of silastic 19 Fr chest tubes were left at the discretion of the operating surgeon.
  Arms: Standard drainage
Device: Active Tube Clearance drainage — One (1) PleuraFlow chest tube must be placed in the anterior mediastinum. The other chest tube(s) may be placed at the discretion of the operator. Chest tubes with internal diameter 28 Fr shall be used. Use of silastic 19 Fr chest tubes were left at the discretion of the operating surgeon.
  Arms: Active Tube Clearance drainage

SUMMARY:
The purpose of this study is to assess the effectiveness of the PleuraFlow® Active Tube Clearance (ATC) technology in reducing the rate of postoperative atrial fibrillation (POAF) among post cardiac surgery patients and to evaluate the impact of Active Tube Clearance (ATC) on other complications, such as retained blood syndrome (RBS), a composite endpoint including re-exploration for bleeding or tamponade, and interventions for hemothorax, pericardial or pleural effusion.

DETAILED DESCRIPTION:
Data will be collected and stored at the department of surgery of Montreal Heart Institute. Only the principal investigator and study coordinators will have access to the database.

The primary analysis will be an intention-to-treat (ITT) analysis comparing the POAF rate in the PleuraFlow® group to the POAF rate in the control group. Based on findings from our institutional clinical database at the Montreal Heart Institute, the local incidence of POAF after cardiac surgery is approximately 25% (control group). The proportion in ATC group (the treatment group) is assumed to be 0,2500 under the null hypothesis and 0,1500 under the alternative hypothesis. Group sample sizes of 254 in each group achieve 80% power to detect a difference between the group proportions of 0,1000 using a Chi-Square test with a significance level of 0.0476. This significance level is computed using the O'Brien-Fleming method and accounts for the interim analysis that is planned after 300 randomized subjects have completed their 30-day follow-up.

POAF and intervention to treat RBS rates and all other categorical event rates will be compared using chi-square tests. Multiple logistic regressions to adjust for potential confounding factors will also be used. Odds ratio and associated 95% confidence intervals will be computed for descriptive purpose. Goodness of fit will be checked using Hosmer-Lemeshow statistics. Quantitative endpoints will be investigated using Student t-tests. Analysis of covariance may also be used to account for potential confounding factors. Nonparametric tests or data transformation may be used if quantitative endpoints are not normally distributed. Correlations and associated 95% confidence intervals will be computed for descriptive purpose. An interim analysis will be conducted on the first 300 randomized subjects completing their 30-day follow-up. The primary endpoint (POAF rate) will be compared between the PleuraFlow® group and the control group using a chi-square test. The significance level for this test will be 0.0076, as computed using the O'Brien-Fleming method. If the p-value of the chi-square test is below this bound at the interim analysis, the study will be stopped for efficacy. Otherwise, the study will continue up to the planned 508 patients. As a result of this interim look, the final analysis of the primary endpoint would require a p < 0.0476 to be declared statistically significant. Analysis of the secondary endpoints and other outcomes will be conducted at the 0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

1. Admission for coronary artery bypass graft (CABG), valve replacement or valve repair surgery, or a combination of these surgeries;
2. Surgical procedure(s) on the ascending aorta and/or aortic arch that do not require deep hypothermic arrest (deep hypothermic arrest is defined as < 18° C);
3. Must be in sinus rhythm (SR) for a minimum of 30 days prior to the index surgery and at the start of the index surgery. No patient with history of atrial fibrillation.
4. Sign the institutional review board/institutional ethics committee approved informed consent form after the nature of the study has been explained and questions/concern have been addressed.

Exclusion Criteria:

1. Admitted for surgical treatment of arrhythmia or Atrial fibrillation history;
2. Admitted for cardiac surgery requiring implantation/explantation of a Ventricular Assist Device (VAD) or heart transplant;
3. Admitted for Transcatheter aortic valve replacement (TAVR);
4. Cardiac surgical procedure that requires deep hypothermic arrest (as defined above);
5. New or active endocarditis or myocarditis that is not adequately controlled with medication and/or requires surgical intervention;
6. Documented inherited bleeding disorder(s);or
7. History or known allergies to the device materials.
8. Intervention carried out by a non-participating surgeon

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2015-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Demers, MD MSc, Principal Investigator — Montreal Heart Institute
Locations (2):
- Canada (2):
  - Montreal Heart Institute, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] St-Onge S, Chauvette V, Hamad R, Bouchard D, Jeanmart H, Lamarche Y, Perrault LP, Demers P. Active clearance vs conventional management of chest tubes after cardiac surgery: a randomized controlled study. J Cardiothorac Surg. 2021 Mar 23;16(1):44. doi: 10.1186/s13019-021-01414-0. PMID 33757537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 257 patients were randomized in the Active Tube Clearance (ATC) group for 263 in the standard drainage group prior to early dropouts. Respectively, 241 and 249 patients were followed for the duration of the trial. 100 random patients were included in the direct visual analysis: 57 and 43 in each respective group.
Pre-assignment Details: 30 patients were excluded after randomization because of the identification of an exclusion criteria
  Atrial fibrillation history (n = 10) Transcatheter aortic valve replacement (n = 1) Deep hypothermic arrest (n = 1) Active endocarditis (n = 3) Inherited bleeding disorder (n = 1) Minimally invasive procedure (n = 14)
Groups:
- Active Tube Clearance Drainage: The test arm consists of consecutively enrolled cardiac surgery patients receiving one (1) chest tube using active tube clearance (PleuraFlow®) in the mediastinum and at most three (3) other commercially available standard or silastic chest tubes in the mediastinal, right or left pleural space.
  Active Clearance Technology drainage: One (1) PleuraFlow chest tube must be placed in the anterior mediastinum. The other chest tube(s) may be placed at the discretion of the operator. Chest tubes with internal diameter 28 Fr shall be used. Use of silastic 19 Fr chest tubes were left at the discretion of the operating surgeon.
Period: Overall Study
Arm/Group | Standard Drainage | Active Tube Clearance Drainage
Started | 249 | 241
Completed | 240 | 230
Not Completed | 9 | 11
Not completed — Lost to Follow-up | 9 | 11

BASELINE CHARACTERISTICS:
Groups:
- Standard Drainage: The control arm consist of consecutively enrolled cardiac surgery patients receiving one standard chest tube in the mediastinum and at most three (3) commercially available standard or silastic chest tubes in the mediastinal, right or left pleural space.
  Standard drainage: One (1) chest tube must be placed in the anterior mediastinum. The other chest tube(s) may be placed at the discretion of the operator. Chest tubes with internal diameter 28 French (FR) shall be used. Use of silastic 19F chest tubes were left at the discretion of the operating surgeon.
- Active Tube Clearance Drainage: The test arm consists of consecutively enrolled cardiac surgery patients receiving one (1) chest tube using active tube clearance (PleuraFlow®) in the mediastinum and at most three (3) other commercially available standard or silastic chest tubes in the mediastinal, right or left pleural space.
  Active Clearance Technology drainage: One (1) PleuraFlow chest tube must be placed in the anterior mediastinum. The other chest tube(s) may be placed at the discretion of the operator. Chest tubes with internal diameter 28 FR shall be used. Use of silastic 19F chest tubes were left at the discretion of the operating surgeon.
- Total: Total of all reporting groups
Arm/Group | Standard Drainage | Active Tube Clearance Drainage | Total
Number analyzed (Participants) | 249 | 241 | 490
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (10.8) | 66.8 (8.3) | 66.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 46 | 99
  Male | 196 | 195 | 391
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Atrial Fibrillation
Description: Rate of any episode of new onset of Postoperative Atrial Fibrillation (POAF) in the study group. POAF is defined as any atrial fibrillation episode ≥ 60 min on telemetry or EKG. At any time between post index surgery through hospital discharge.
Time Frame: From post index surgery through hospital discharge, an average of 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Standard Drainage: The control arm consist of consecutively enrolled cardiac surgery patients receiving one (1) standard chest tube in the mediastinum and at most three (3) commercially available standard or silastic chest tubes in the mediastinal, right or left pleural space.
  Standard drainage: One (1) chest tube must be placed in the anterior mediastinum. The other chest tube(s) may be placed at the discretion of the operator. Chest tubes with internal diameter 28 French (Fr) shall be used. Use of silastic 19 Fr chest tubes were left at the discretion of the operating surgeon.
Arm/Group | Standard Drainage | Active Tube Clearance Drainage
Number analyzed (Participants) | 249 | 241
Participants | 39 | 33

2. Secondary Outcome: Number of Participants Requiring Invasive Procedure for Intrathoracic Fluid Removal (Retained Blood Complications)
Description: Any of the following:
  * Re-exploration for bleeding or cardiac tamponade
  * Pericardial drainage procedure (pericardiocentesis or pericardial window)
  * Pleural drainage procedure (thoracentesis, new chest tube, thoracoscopy or lateral thoracotomy)
Time Frame: Within 30 days post index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Drainage | Active Tube Clearance Drainage
Number analyzed (Participants) | 249 | 241
Participants | 27 | 15

3. Secondary Outcome: Number of Participants Requiring Re-exploration for Bleeding or Tamponade
Description: Rate of re-exploration for bleeding or tamponade within 30-day post index surgery
Time Frame: within 30-day post index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Drainage | Active Tube Clearance Drainage
Number analyzed (Participants) | 249 | 241
Participants | 14 | 4

4. Secondary Outcome: Number of Participants Presenting With a Chest Tube Occlusion
Description: Visual observation of mediastinal chest tube lumen upon removal to determine whether it is:
  * patent
  * partially occluded
  * totally occluded
Time Frame: At chest tube removal
Population: 100 random patients were included in this analysis where the chest tubes were visually inspected upon removal by a blinded investigator. They were selected by convenience, when the investigator was available.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Drainage | Active Tube Clearance Drainage
Number analyzed (Participants) | 43 | 57
Participants
  Patent | 26 | 42
  Partially obstructed | 9 | 14
  Totally obstructed | 8 | 1

5. Secondary Outcome: Number of Patients Requiring Pericardial Drainage Procedure
Description: Rate of invasive pericardial drainage procedure within 30-day post index surgery
Time Frame: within 30-day post index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Drainage | Active Tube Clearance Drainage
Number analyzed (Participants) | 249 | 241
Participants | 5 | 2

6. Secondary Outcome: Number of Patients Requiring Pleural Drainage Procedure
Description: Rate of invasive pleural drainage procedure within 30-day post index surgery
Time Frame: within 30-day post index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Drainage | Active Tube Clearance Drainage
Number analyzed (Participants) | 249 | 241
Participants | 8 | 9

7. Other Pre Specified Outcome: Number of Patients Being Readmitted
Description: Frequency of readmission for any indication
Time Frame: Within 30 days post index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Drainage | Active Tube Clearance Drainage
Number analyzed (Participants) | 249 | 241
Participants | 24 | 27

8. Other Pre Specified Outcome: Total Chest Tube Output
Description: Total chest tube output (milliliter)
Time Frame: At chest tube removal
Measure: Median (95% Confidence Interval); unit: milliliters
Arm/Group | Standard Drainage | Active Tube Clearance Drainage
Number analyzed (Participants) | 249 | 241
milliliters | 640 [430 to 815] | 580 [440 to 900]

ADVERSE EVENTS:
Time Frame: within 30-day post index surgery
Groups:
- Standard Drainage: The control arm consist of consecutively enrolled cardiac surgery patients receiving one (1) standard chest tube in the mediastinum and at most three (3) commercially available standard or silastic chest tubes in the mediastinal, right or left pleural space.
  Standard drainage: One (1) chest tube must be placed in the anterior mediastinum. The other chest tube(s) may be placed at the discretion of the operator. Chest tubes with internal diameter 28 French (Fr) shall be used. Use of silastic 19Fr chest tubes were left at the discretion of the operating surgeon.
- Active Tube Clearance Drainage: The test arm consists of consecutively enrolled cardiac surgery patients receiving one (1) chest tube using active tube clearance (PleuraFlow®) in the mediastinum and at most three (3) other commercially available standard or silastic chest tubes in the mediastinal, right or left pleural space.
  Active Tube Clearance drainage: One (1) PleuraFlow chest tube must be placed in the anterior mediastinum. The other chest tube(s) may be placed at the discretion of the operator. Chest tubes with internal diameter 28 Fr shall be used. Use of silastic 19Fr chest tubes were left at the discretion of the operating surgeon.
Arm/Group | Standard Drainage | Active Tube Clearance Drainage
All-Cause Mortality (participants affected / at risk) | 4/240 | 3/230
Serious Adverse Events (participants affected / at risk) | 0/240 | 0/230
Other Adverse Events (participants affected / at risk) | 0/230 | 0/240

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT02808897/Prot_SAP_000.pdf